CLINICAL TRIAL: NCT00601965
Title: CBT Augmentation of SSRI Treatment for Geriatric GAD
Brief Title: Antidepressant Treatment Plus Cognitive Behavioral Therapy for Generalized Anxiety Disorder in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34MH080151 (NIH); R34MH080151 (NIH); NCT00601965 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Escitalopram; Sugars; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CBT/Escitalopram (Experimental): 12 weeks open-label escitalopram (10-20mg/day as tolerated), followed by 16 weeks individual cognitive behavioral therapy plus continuation escitalopram at same dose as end of first 12 weeks, followed by 28 weeks maintenance escitalopram at same dose as at end of first 12 weeks. Up to 3 booster sessions of CBT allowed during the 28 week maintenance phase. CBT consists of 16 sessions of relaxation training, cognitive restructuring, and problem-solving skills training.
  Interventions: Drug: Escitalopram; Behavioral: Cognitive behavioral therapy (CBT)
- No CBT/escitalopram (Active Comparator): 12 weeks open-label escitalopram (10-20 mg/day as tolerated), followed by 16 weeks continuation escitalopram at same dose as at end of first 12 weeks, followed by 28 weeks maintenance escitalopram at same dose as at end of first 12 weeks.
  Interventions: Drug: Escitalopram
- CBT/placebo (Placebo Comparator): 12 weeks open-label escitalopram (10-20mg/day as tolerated), followed by 16 weeks individual cognitive behavioral therapy plus continuation escitalopram at same dose as end of first 12 weeks, followed by 28 weeks of pill placebo. 28 weeks of pill placebo includes a taper period of a duration dependent on the initial dose of escitalopram, but in all cases taper to placebo is complete after 8 weeks. Up to 3 booster sessions of CBT allowed during the 28 week maintenance phase. CBT consists of 16 sessions of relaxation training, cognitive restructuring, and problem-solving skills training.
  Interventions: Drug: Placebo; Behavioral: Cognitive behavioral therapy (CBT)
- No CBT/placebo (Placebo Comparator): 12 weeks open-label escitalopram, 16 weeks continuation escitalopram, 28 weeks pill placebo
  12 weeks open-label escitalopram (10-20 mg/day as tolerated), followed by 16 weeks continuation escitalopram at same dose as at end of first 12 weeks, followed by 28 weeks of pill placebo. 28 weeks of pill placebo includes a taper period of a duration dependent on the initial dose of escitalopram, but in all cases taper to placebo is complete after 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 20 mg daily oral escitalopram
  Other Names: Lexapro
  Arms: CBT/Escitalopram; No CBT/escitalopram
Drug: Placebo — Placebo pill of daily oral escitalopram
  Other Names: Sugar pill
  Arms: CBT/placebo; No CBT/placebo
Behavioral: Cognitive behavioral therapy (CBT) — 16 weekly 1-hour sessions
  Other Names: CBT
  Arms: CBT/Escitalopram; CBT/placebo

SUMMARY:
This study will assess whether adding cognitive behavioral therapy to the antidepressant escitalopram is effective in reducing anxiety in older adults with generalized anxiety disorder.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) affects nearly 6.8 million adults in the United States. GAD is diagnosed when a person spends at least 6 months excessively worrying over everyday problems to the point that carrying out normal life becomes difficult. People with GAD face each day with intense anxiety and tension and are unable to alleviate their worries. Physical symptoms of GAD include muscle aches, nausea, sweating, exhaustion, irritability, frequent urination, shaking, and hot flashes. People with GAD often experience other anxiety disorders, depression, or substance abuse, all of which can worsen symptoms of GAD. This makes early and appropriate treatment for GAD important. Current treatments for GAD include medication and/or types of psychotherapy. This study will assess whether adding cognitive behavioral therapy (CBT) to the antidepressant escitalopram is effective in reducing anxiety in older adults with GAD.

Participation in this double-blind study will last up to 13 months. Participants will be asked to stop any current treatments for anxiety or depression for the duration of the study. Participants will begin taking one pill of the medication escitalopram daily for 12 weeks. Dosage will be increased to two pills each day if symptoms do not improve within 4 weeks. After 12 weeks, all participants will continue taking escitalopram for an additional 16 weeks. In addition, some participants will be randomly assigned to receive 16 weekly sessions of CBT, lasting 1 hour each. CBT sessions will involve learning relaxation techniques and other skills to manage anxiety and completing 30-minute at-home practice assignments each day. A family member will accompany participants to the first four CBT sessions. All participants will be asked to provide information for a close contact, who will be interviewed at baseline, Month 3, and Month 7 about how the participant's anxiety is affecting his or her relationships.

After the 16-week period, participants will again be randomly assigned to receive either continued escitalopram or a placebo for an additional 28 weeks. Participants assigned to the placebo will be gradually tapered off escitalopram over a 6-week period. Participants who were receiving CBT will receive three more sessions. Throughout the study, participants will be asked to complete various assessments, including questionnaires, memory and thinking tests, and attention evaluations. Blood samples will be taken at Weeks 2 and 8, and saliva samples will be taken at baseline and Weeks 12, 28, and 56.

ELIGIBILITY:
Inclusion Criteria:

* Principal (i.e., most severe or pressing problem) or co-principal current diagnosis of generalized anxiety disorder
* Pretreatment score of at least 17 on Hamilton Anxiety Rating Scale

Exclusion Criteria:

* Principal diagnosis other than GAD
* Clinically judged too psychiatrically unstable to participate in the study
* Cognitive impairment or dementia
* Alcohol or other substance use disorder within 6 months prior to study entry
* Lifetime diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, or bipolar disorder
* Serious, unstable, or terminal medical condition that would compromise study participation or preclude the use of escitalopram, as determined by a review of medical records
* Use of psychotropics that could not be safely tapered and discontinued for at least 2 weeks prior to study entry
* Use of depot neuroleptics within 6 weeks prior to study entry
* Unwillingness to terminate other forms of psychotherapy
* Already received adequate trial of escitalopram or CBT

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L. Wetherell, PhD, Principal Investigator — UCSD and VMRF/VASDHS
Locations (3):
- United States (3):
  - UCSD Outpatient Psychiatric Services, San Diego, California
  - Washington University, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wetherell JL, Petkus AJ, White KS, Nguyen H, Kornblith S, Andreescu C, Zisook S, Lenze EJ. Antidepressant medication augmented with cognitive-behavioral therapy for generalized anxiety disorder in older adults. Am J Psychiatry. 2013 Jul;170(7):782-9. doi: 10.1176/appi.ajp.2013.12081104. PMID 23680817

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram + CBT: 12 weeks open-label escitalopram, 16 weeks cognitive behavioral therapy plus continuation escitalopram, 28 weeks maintenance escitalopram
  Escitalopram: 20 mg daily oral escitalopram
  Cognitive behavioral therapy (CBT): 16 weekly 1-hour sessions
- Escitalopram + no CBT: 12 weeks open-label escitalopram, 16 weeks continuation escitalopram, 28 weeks maintenance escitalopram
  Escitalopram: 20 mg daily oral escitalopram
- Placebo + CBT: 12 weeks open-label escitalopram, 16 weeks cognitive behavioral therapy plus continuation escitalopram, 28 weeks pill placebo
  Escitalopram: 20 mg daily oral escitalopram
  Placebo: Placebo pill of daily oral escitalopram
  Cognitive behavioral therapy (CBT): 16 weekly 1-hour sessions
- Placebo + no CBT: 12 weeks open-label escitalopram, 16 weeks continuation escitalopram, 28 weeks pill placebo
  Escitalopram: 20 mg daily oral escitalopram
  Placebo: Placebo pill of daily oral escitalopram
Period: Overall Study
Arm/Group | Escitalopram + CBT | Escitalopram + no CBT | Placebo + CBT | Placebo + no CBT
Started | 18 | 18 | 19 | 18
Completed | 18 | 16 | 19 | 17
Not Completed | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: please see Wetherell et al. (2013), Antidepressant Medication Augmented with Cognitive-Behavioral Therapy for Generalized Anxiety Disorder in Older Adults, American Journal of Psychiatry, 170:782-9.
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram + CBT | Escitalopram + no CBT | Placebo + CBT | Placebo + no CBT | Total
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.7) | 70.3 (8.6) | 70.2 (8.1) | 66.9 (5.7) | 69.5 (7.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 8 | 6 | 27
  >=65 years | 12 | 11 | 11 | 12 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 13 | 13 | 52
  Male | 6 | 4 | 6 | 5 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13 | 13 | 16 | 15 | 57
  Hispanic | 1 | 1 | 1 | 2 | 5
  African American | 4 | 4 | 1 | 1 | 10
  Other | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 19 | 18 | 73

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale is a clinician-rated measure of cognitive and somatic anxiety symptoms. It consists of 14 items, each of which is scored on a 0-4 scale, summed for a total score ranging from 0 to 56. Inclusion criteria for this study included a Hamilton score >= 17. The Hamilton, administered by blind raters, will be used to test hypotheses number 1 and 2. The outcome of interest is the number of participants who relapse, defined as having a Hamilton increase of >=5, for a total Hamilton >=14, relative to the end of the continuation phase (week 28), for a duration of at least 2 weeks, plus both clinician's and participant's judgment that the participant is experiencing a recurrence of anxiety symptoms. HAMA scores range from 0 (no anxiety) to 56 (high anxiety).
Time Frame: 56 weeks
Measure: Number; unit: participants
Arm/Group | Escitalopram + CBT | Escitalopram + no CBT | Placebo + CBT | Placebo + no CBT
Number analyzed (Participants) | 18 | 16 | 19 | 17
participants | 18 | 15 | 14 | 8
Statistical Analysis 1: Comparison: Escitalopram + CBT vs Escitalopram + no CBT vs Placebo + CBT vs Placebo + no CBT; Test type: Superiority or Other; p < .001, Log Rank; Log rank test = 32.67, df = 3

2. Primary Outcome: Penn State Worry Questionnaire
Description: The Penn State Worry Questionnaire is a 16-item measure of pathological worry. Scores range from 16-80, with higher scores indicating higher levels of worry.
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram + CBT | Escitalopram + no CBT | Placebo + CBT | Placebo + no CBT
Number analyzed (Participants) | 18 | 19 | 18 | 18
units on a scale | 52.8 (2.6) | 53.4 (10.3) | 54.4 (11.7) | 57.7 (12.7)
Statistical Analysis 1: Comparison: Escitalopram + CBT vs Escitalopram + no CBT vs Placebo + CBT vs Placebo + no CBT; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; Beta = -0.48, 95% CI = -0.84 to -0.11

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Escitalopram + CBT | Escitalopram + no CBT | Placebo + CBT | Placebo + no CBT
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No